CLINICAL TRIAL: NCT02593318
Title: Trial of Oxaloacetate in Alzheimer's Disease (TOAD)
Acronym: TOAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Russell Swerdlow (Other)
Responsible Party: Sponsor-Investigator, Russell Swerdlow, Gene and Marge Sweeney Professor of Neurology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002242
Record Dates: First submitted 2015-10-08; First posted 2015-11-02 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer's Disease (AD)
Keywords: energy metabolism; oxaloacetate
MeSH Terms: conditions — Alzheimer Disease | interventions — Oxaloacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 - Oxaloacetate (OAA) 1 gram/day (Experimental): Participants take 1 gram of OAA per day for period of 4 weeks
  Interventions: Drug: Oxaloacetate (OAA) 1g
- Part 2 - Oxaloacetate (OAA)2 gram/day (Experimental): Participants take 2 grams of OAA per day for period of 4 weeks
  Interventions: Drug: Oxaloacetate (OAA) 2g

INTERVENTIONS:
Drug: Oxaloacetate (OAA) 1g — Pills to be taken orally in 500mg dose two times per day
  Other Names: Oxobutanedioic acid; Oxaloacetic acid; Oxalacetic acid; 2-Oxosuccinic acid; Ketosuccinic acid
  Arms: Part 1 - Oxaloacetate (OAA) 1 gram/day
Drug: Oxaloacetate (OAA) 2g — Pills to be taken orally in 1000mg dose two times per day.
  Other Names: Oxobutanedioic acid; Oxaloacetic acid; Oxalacetic acid; 2-Oxosuccinic acid; Ketosuccinic acid
  Arms: Part 2 - Oxaloacetate (OAA)2 gram/day

SUMMARY:
The purpose of this study is to determine if oxaloacetate (OAA) is safe and tolerable at doses of up to 2 grams per day in people with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive brain disorder that causes memory and thinking problems. The exact cause of AD is unknown. Researchers believe mitochondria (the part of your cells that produce energy) might be linked to symptoms of AD. Some studies have shown that the brains in patients with Alzheimer's disease have reduced mitochondrial activity, have fewer mitochondria present in the nerve cells, and have reduced ability to utilize glucose (sugar) for energy.

Oxaloacetate (OAA) is a natural chemical that has been shown to have an effect on brain mitochondrial activity and brain energy in non-human animals.

This study is divided into two parts. In the first part of the study, researchers will test whether a dose of 1 gram per day of OAA, taken for approximately 4 weeks in 15 people with AD is safe and tolerable. After all 15 participants in part 1 have completed their participation, and it is determined that the study drug was safe at this dose, the second part of the study will begin. In part 2, researchers will test a dose of 2 grams per day of OAA, taken for approximately 4 weeks in 15 people with AD, to assess safety at this dose.

Participants will be in this study for about 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of probable Alzheimer's disease (AD) per McKhann et al. criteria [9];
* Have a clinical dementia rating (CDR) score of 0.5 or 1 at time of their last University of Kansas Alzheimer's Disease Center (KU ADC) assessment;
* Have a Mini Mental Status Exam (MMSE) score of 15-28 at the TOAD screening visit;
* Have a reliable and competent study partner who is willing to accompany the participant to all study visits, monitor compliance of study medication administration, and observe/report any changes in the participant's health throughout the study duration;
* Are on stable doses of concurrent medications for at least 4 weeks prior to the TOAD screening visit; and
* Speaks English as his/her primary language.
* If female of child-bearing potential, must have a negative urine pregnancy test at TOAD screening visit (and must agree to use of contraception throughout the trial)

Exclusion Criteria:

* Dementia due to causes other than AD;
* Potentially confounding, serious, or unstable medical conditions such as:

  * insulin-dependent diabetes mellitus
  * cancer within the past 3 years (except basal cell, squamous cell, or localized prostate cancer)
  * a recent cardiac event (i.e. heart attack, angioplasty, etc. within the 6 months prior to screening visit)
  * other conditions that pose a potential safety risk or confounding factor in the investigator's opinion;
* Any abnormal physical examination assessment or vital sign assessment at TOAD screening visit that is deemed to be clinically significant by the principal investigator;
* Any abnormal clinical laboratory test result at TOAD screening visit that is deemed to be clinically significant by the principal investigator.
* Any contraindication for undergoing magnetic resonance spectroscopy (MRS), such as the presence of metal implants, a cardiac pacemaker that is not compatible with MRS, or severe claustrophobia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Swerdlow, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Original plan was to enroll 30 participants. After enrolling 30 participants, two enrolled participants were withdrawn from the study after assignment to groups but did not complete post treatment data collection. Therefore those two were replaced so that total number of participants who completed post treatment data was 30, increasing the total number of enrolled participants to 32.
Groups:
- Part 1 - Oxaloacetate (OAA) 1 Gram/Day: Participants take 1 gram of OAA per day for period of 4 weeks
  Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study
- Part 2 - Oxaloacetate (OAA)2 Gram/Day: Participants take 2 grams of OAA per day for period of 4 weeks
  Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study
Period: Overall Study
Arm/Group | Part 1 - Oxaloacetate (OAA) 1 Gram/Day | Part 2 - Oxaloacetate (OAA)2 Gram/Day
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Oxaloacetate (OAA) 1 Gram/Day | Part 2 - Oxaloacetate (OAA)2 Gram/Day | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (5.7) | 71.3 (8.1) | 70.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Baseline MMSE [Mean (Standard Deviation); unit: Scores on a Scale] — The Mini-Mental State Exam (MMSE) is a 30 point questionnaire that measures cognitive impairment. Score ranges from 0 to 30 and are adjusted based on education level of the participant. A score of 20 to 24 suggests mild dementia, a score of 13 to 20 suggest moderate dementia, and a score of 12 or less suggests severe dementia.
  Scores on a Scale | 21.5 (4.3) | 21.9 (3.2) | 21.7 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicity Events
Description: The number of dose limiting toxicity events will be determined by change in safety labs, physical and neurological exams, vital signs, cognitive measures, signs and symptoms.
Time Frame: Change from Baseline to Week 4
Measure: Number; unit: Dose Limiting Toxicity Events
Arm/Group | Part 1 - Oxaloacetate (OAA) 1 Gram/Day | Part 2 - Oxaloacetate (OAA)2 Gram/Day
Number analyzed (Participants) | 15 | 15
Dose Limiting Toxicity Events | 0 | 0

2. Secondary Outcome: Change in Brain Glucose Metabolic Rate as Determined by Fluorodeoxyglucose Positron Emission Tomography (FDG PET)
Description: Fluorodeoxyglucose positron emission tomography (FDG PET)
Time Frame: Change from Baseline to Week 4
Reporting Status: Not Posted

3. Secondary Outcome: Change in Brain Lactate Levels as Determined by Magnetic Resonance Spectroscopy (MRS)
Description: magnetic resonance spectroscopy (MRS)
Time Frame: Change from Baseline to Week 4
Reporting Status: Not Posted

4. Secondary Outcome: Plasma Levels in 500 mg Bid Cohort at Baseline, 60 and 90 Minutes Post-Dose
Description: For the 1 g/ day (500 mg bid) cohort, baseline blood sample will be obtained just before 500 mg OAA is administered. Blood samples to be drawn again at 60 min and 90 min post administration of dose. The amount of OOA in the blood will be measured at each of the three time points.
Time Frame: Change from dose to 60 min post dose and 90 min post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1 - Oxaloacetate (OAA) 1 Gram/Day - Baseline: Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Baseline blood sample obtained prior to 500 mg OOA administered
- Part 1 - Oxaloacetate (OAA) 1 Gram/Day - 60 Minutes Post Administration of Dose: Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Baseline blood sample drawn 60 minutes post administration of dose.
- Part 1 - Oxaloacetate (OAA) 1 Gram/Day - 90 Minutes Post Administration of Dose: Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Blood sample drawn 90 minutes post administration of dose.
Arm/Group | Part 1 - Oxaloacetate (OAA) 1 Gram/Day - Baseline | Part 1 - Oxaloacetate (OAA) 1 Gram/Day - 60 Minutes Post Administration of Dose | Part 1 - Oxaloacetate (OAA) 1 Gram/Day - 90 Minutes Post Administration of Dose
Number analyzed (Participants) | 15 | 15 | 15
ng/mL | 94 (102) | 63 (55) | 87 (80)

5. Secondary Outcome: Plasma Levels in 1000 mg Bid Cohort at Baseline, 60 and 90 Minutes Post-Dose
Description: For the 2 g/ day (1000 mg bid) cohort, baseline blood sample will be obtained before 1000 mg OAA is administered. Blood samples to be drawn again at 60 min and 90 min post administration of dose. Plasma levels of OOA will be measured at each of the three timepoints.
Time Frame: Change from dose to 60 min post dose and 90 min post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Oxaloacetate (OAA) 2 Gram/Day - Baseline Blood Sample: Participants take 2 gram of OAA per day for period of 4 weeks
  Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Blood sample drawn at baseline prior to dose administration.
- Oxaloacetate (OAA)2 Gram/Day - 60 Minutes Post Administration: Participants take 2 grams of OAA per day for period of 4 weeks
  Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Blood sample drawn at 60 minutes post administration of dose.
- Oxaloacetate (OAA)2 Gram/Day - 90 Minutes Post Administration of Dose: Participants take 2 grams of OAA per day for period of 4 weeks
  Oxaloacetate (OAA): Pills to be taken orally in 500mg or 1000mg doses two times per day depending on the part of the study. Blood sample to be drawn 90 minutes post administration of dose
Arm/Group | Oxaloacetate (OAA) 2 Gram/Day - Baseline Blood Sample | Oxaloacetate (OAA)2 Gram/Day - 60 Minutes Post Administration | Oxaloacetate (OAA)2 Gram/Day - 90 Minutes Post Administration of Dose
Number analyzed (Participants) | 15 | 15 | 15
ng/mL | 1400 (962) | 1355 (690) | 1363 (759)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Part 1 - Oxaloacetate (OAA) 1 Gram/Day | Part 2 - Oxaloacetate (OAA)2 Gram/Day
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Oxaloacetate (OAA) 1 Gram/Day (N=15) | Part 2 - Oxaloacetate (OAA)2 Gram/Day (N=15)
Increased confusion (Nervous system disorders) | 2 (2) | 0 (0)
Cervical Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Breast calcification (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT02593318/Prot_000.pdf